CLINICAL TRIAL: NCT02496923
Title: A Randomised Controlled Trial of High-flow Nasal Oxygen (Optiflow™) and Standard Oxygen Therapy in High-risk Patients After Cardiac Surgery
Brief Title: High Flow Nasal Oxygen Therapy (Optiflow™) in High-risk Cardiac Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P2043
Record Dates: First submitted 2015-06-22; First posted 2015-07-14 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Cardiac Surgery
Keywords: prophylactic NHFO; risk of developing postoperative pulmonary complications; reduces hospital length of stay

ARMS (2):
- High flow nasal oxygen therapy (Optiflow™) (Experimental): In patients randomised to receive high flow nasal oxygen therapy (HFNO) the gas flow through the HFNO will be calculated for each patient, based on their body characteristics, and comfort level. The standard starting flow rate will be 30 L/min, and this will be adjusted up or down between a range of 20-50 L/min with the aim of achieving both patient comfort and a respiratory rate of less than 16 breaths per minute.
  Interventions: Device: High flow nasal oxygen therapy (Optiflow™)
- Standard oxygen therapy (Hudson face mask or nasal prongs) (Active Comparator): Patients randomised to receive standard oxygen therapy will be fitted with a soft face mask or nasal prongs, and the oxygen flow titrated to provide pulse oxygen saturation of at least 95% (93% for those at risk of hypercapnic respiratory failure such as confirmed COPD patients and morbidly obese patients). The standard oxygen therapy group will have their oxygen gas flow reduced to the minimum level which provides saturations of at least 95% (93% for those at risk of hypercapnic respiratory failure such as patients with confirmed COPD and morbidly obese patients).
  Interventions: Device: Standard oxygen therapy (Hudson Type face mask or nasal prongs)

INTERVENTIONS:
Device: High flow nasal oxygen therapy (Optiflow™)
  Other Names: (Optiflow™)
  Arms: High flow nasal oxygen therapy (Optiflow™)
Device: Standard oxygen therapy (Hudson Type face mask or nasal prongs)
  Other Names: Hudson Type face mask
  Arms: Standard oxygen therapy (Hudson face mask or nasal prongs)

SUMMARY:
Background:

High risk patients with lung disease who undergo cardiac surgery are at significant risk of postoperative complications leading to prolonged hospital stay. One method of reducing the risk of lung complications is to treat patients with non-invasive ventilation or continuous positive airways pressure postoperatively. However, this often requires admission to a high dependency unit or intensive care, and is uncomfortable because of the need for a tight fitting mask, as well as being labour intensive and costly. Nasal high flow oxygen (Optiflow™) is a new alternative as it provides warmed humidified oxygen at high flow, and also has been shown to assist breathing and improve recovery. It is comfortable during use and indeed may be more comfortable than standard (dry) oxygen via a facemask (Hudson type) or nasal prongs. It may be administered on a normal ward, however its routine use in high risk patients with lung conditions such as asthma, chronic obstructive pulmonary disease, recent chest infections and heavy smokers has not been tested before.

Aims/Objectives:

The primary aim of this clinical trial is to determine if prophylactic nasal high flow oxygen (Optiflow™) therapy in cardiac surgical patients at high-risk of developing post-operative pulmonary complications is associated with shorter hospital length of stay.

Methods:

High risk adult patients who are scheduled to undergo cardiac surgery will be recruited with full ethical approval and informed consent. Before surgery, each patient will perform a 6- minute walking test under the supervision of a physiotherapist. This simple tests measures how far patients can walk in 6 minutes. Additionally, patients will undergo spirometry testing which is used to assess how well the lungs work by measuring how much air the patient inhales and exhales and how quickly they exhale. Patients will thereafter undergo surgery under general anaesthesia as they would normally. After the operation they will be looked after following our recovery protocols, incorporating pain relief, regular physiotherapy, early mobilisation and eating and drinking, and removal of chest drains and tubes as soon as possible.

On arrival in the critical care area after their surgery, patients will be randomly assigned to receive supplemental oxygen via a soft facemask (Hudson Type) (standard group), or via high-flow nasal cannulae(Optiflow™) (intervention group). Patients will be administered oxygen for at least 24 hours after surgery.

Patients who develop breathing difficulty will receive treatment based on their clinical need. On the fifth or sixth postoperative day they will repeat the walking test and spirometry. The investigators will use a short questionnaire to determine if there is any difference in how patients feel they recovered before they leave hospital and how quickly they returned to normal activities after discharge, and also to evaluate how they tolerated either the facemask (Hudson Type) or high flow nasal cannulae (Optiflow™).

The investigators have used data from previous studies to calculate that a total of 74 patients will be needed to take part, in order to evaluate whether high flow nasal oxygen (Optiflow™) leads to reduced length of hospital stay after high risk cardiac surgery compared with usual care oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for inclusion if:

* they are aged over 18 years
* are undergoing elective cardiac surgery (coronary artery bypass grafting, valve surgery or both)
* they have one or more patient-related risk factor for post-operative pulmonary complications (COPD, asthma, lower respiratory tract infection in last 4 weeks, body mass index≥35 kg/m2 current (last 6 weeks) heavy smokers (> 10 packyears)).
* they are capable of performing a 6MWT - The 6MWT is a clinical exercise test, and is popular in clinical practice because it aids clinical decision making, and because of the belief that it provides a better estimate of functional capacity than resting cardiorespiratory measurements (24). The 6MWT is the most popular clinical exercise test, which is used for postoperative evaluation after lung surgery and has also been validated in cardiac surgery

Exclusion Criteria:

* Contraindication to high flow nasal oxygen such as nasal septal defect.
* Not met extubation criteria by 10am the day after surgery (Day 1).
* Need for CPAP pre-operatively.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay (days) | 10 days (plus or minus 3 days) after surgery
  To determine if prophylactic nasal high flow oxygen (NHFO) therapy in cardiac surgical patients at high-risk of developing post-operative pulmonary complications, is associated with shorter hospital length of stay (days).

SECONDARY OUTCOMES:
Early postoperative recovery | 1 month
  Early postoperative recovery, as determined by performance on a 6 minute walking test, compared with patients who receive standard (soft face mask or nasal prongs) oxygen therapy
Early postoperative lung function | Approximately 1 week after surgery
  Early postoperative lung function, tested by spirometry
Intensive care unit readmission rate | First 24 hours after surgery
  Determine if prophylactic NHFO therapy in high-risk cardiac surgical patients, is associated with reduced intensive care unit readmission rate.
Intensive Care Unit length of stay (hours) | 30 hours (plus or minus 24 hours)
  Determine if prophylactic NHFO therapy in high-risk cardiac surgical patients, is associated with shorter ICU length of stay (days).
Escalation of respiratory support | Determine if prophylactic NHFO in high-risk cardiac surgical patients, is associated with reduced requirement for escalation of respiratory support (invasive or non-invasive respiratory support) First 24 hours after surgery
  First 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vasileios Zochios, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge, CB23 3RE, United Kingdom
Locations (1):
- Department of Cardiothoracic Anaesthesia and Critical Care Medicine, Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Background] Pasquina P, Merlani P, Granier JM, Ricou B. Continuous positive airway pressure versus noninvasive pressure support ventilation to treat atelectasis after cardiac surgery. Anesth Analg. 2004 Oct;99(4):1001-1008. doi: 10.1213/01.ANE.0000130621.11024.97. PMID 15385340
- [Background] Wynne R, Botti M. Postoperative pulmonary dysfunction in adults after cardiac surgery with cardiopulmonary bypass: clinical significance and implications for practice. Am J Crit Care. 2004 Sep;13(5):384-93. PMID 15470854
- [Background] Taggart DP, el-Fiky M, Carter R, Bowman A, Wheatley DJ. Respiratory dysfunction after uncomplicated cardiopulmonary bypass. Ann Thorac Surg. 1993 Nov;56(5):1123-8. doi: 10.1016/0003-4975(95)90029-2. PMID 8239811
- [Background] Weissman C. Pulmonary complications after cardiac surgery. Semin Cardiothorac Vasc Anesth. 2004 Sep;8(3):185-211. doi: 10.1177/108925320400800303. PMID 15375480
- [Background] Adabag AS, Wassif HS, Rice K, Mithani S, Johnson D, Bonawitz-Conlin J, Ward HB, McFalls EO, Kuskowski MA, Kelly RF. Preoperative pulmonary function and mortality after cardiac surgery. Am Heart J. 2010 Apr;159(4):691-7. doi: 10.1016/j.ahj.2009.12.039. PMID 20362731
- [Background] Manganas H, Lacasse Y, Bourgeois S, Perron J, Dagenais F, Maltais F. Postoperative outcome after coronary artery bypass grafting in chronic obstructive pulmonary disease. Can Respir J. 2007 Jan-Feb;14(1):19-24. doi: 10.1155/2007/378963. PMID 17315054
- [Background] Leavitt BJ, Ross CS, Spence B, Surgenor SD, Olmstead EM, Clough RA, Charlesworth DC, Kramer RS, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Long-term survival of patients with chronic obstructive pulmonary disease undergoing coronary artery bypass surgery. Circulation. 2006 Jul 4;114(1 Suppl):I430-4. doi: 10.1161/CIRCULATIONAHA.105.000943. PMID 16820614
- [Background] Duggan M, Kavanagh BP. Pulmonary atelectasis: a pathogenic perioperative entity. Anesthesiology. 2005 Apr;102(4):838-54. doi: 10.1097/00000542-200504000-00021. PMID 15791115
- [Background] Lumb AB, Greenhill SJ, Simpson MP, Stewart J. Lung recruitment and positive airway pressure before extubation does not improve oxygenation in the post-anaesthesia care unit: a randomized clinical trial. Br J Anaesth. 2010 May;104(5):643-7. doi: 10.1093/bja/aeq080. Epub 2010 Mar 30. PMID 20354010
- [Background] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Background] Kindgen-Milles D, Muller E, Buhl R, Bohner H, Ritter D, Sandmann W, Tarnow J. Nasal-continuous positive airway pressure reduces pulmonary morbidity and length of hospital stay following thoracoabdominal aortic surgery. Chest. 2005 Aug;128(2):821-8. doi: 10.1378/chest.128.2.821. PMID 16100174
- [Background] Lenique F, Habis M, Lofaso F, Dubois-Rande JL, Harf A, Brochard L. Ventilatory and hemodynamic effects of continuous positive airway pressure in left heart failure. Am J Respir Crit Care Med. 1997 Feb;155(2):500-5. doi: 10.1164/ajrccm.155.2.9032185.
- [Background] Westerlind A, Nilsson F, Ricksten SE. The use of continuous positive airway pressure by face mask and thoracic epidural analgesia after lung transplantation. Gothenburg Lung Transplant Group. J Cardiothorac Vasc Anesth. 1999 Jun;13(3):249-52. doi: 10.1016/s1053-0770(99)90258-6. PMID 10392672
- [Background] Parke RL, Eccleston ML, McGuinness SP. The effects of flow on airway pressure during nasal high-flow oxygen therapy. Respir Care. 2011 Aug;56(8):1151-5. doi: 10.4187/respcare.01106. Epub 2011 Apr 15. PMID 21496369
- [Background] Parke R, McGuinness S, Eccleston M. Nasal high-flow therapy delivers low level positive airway pressure. Br J Anaesth. 2009 Dec;103(6):886-90. doi: 10.1093/bja/aep280. Epub 2009 Oct 20. PMID 19846404
- [Background] Frizzola M, Miller TL, Rodriguez ME, Zhu Y, Rojas J, Hesek A, Stump A, Shaffer TH, Dysart K. High-flow nasal cannula: impact on oxygenation and ventilation in an acute lung injury model. Pediatr Pulmonol. 2011 Jan;46(1):67-74. doi: 10.1002/ppul.21326. Epub 2010 Nov 23. PMID 21171186
- [Background] Cuquemelle E, Lellouche F. Assessment of humidification performance: still no easy method! Respir Care. 2013 Sep;58(9):1559-61. doi: 10.4187/respcare.02761. No abstract available. PMID 23981591
- [Background] Manley BJ, Owen LS, Doyle LW, Andersen CC, Cartwright DW, Pritchard MA, Donath SM, Davis PG. High-flow nasal cannulae in very preterm infants after extubation. N Engl J Med. 2013 Oct 10;369(15):1425-33. doi: 10.1056/NEJMoa1300071. PMID 24106935
- [Background] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Background] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Background] Corley A, Bull T, Spooner AJ, Barnett AG, Fraser JF. Direct extubation onto high-flow nasal cannulae post-cardiac surgery versus standard treatment in patients with a BMI >/=30: a randomised controlled trial. Intensive Care Med. 2015 May;41(5):887-94. doi: 10.1007/s00134-015-3765-6. Epub 2015 Apr 8. PMID 25851385
- [Background] Weisman IM, Zeballos RJ. Clinical exercise testing. Clin Chest Med. 2001 Dec;22(4):679-701, viii. doi: 10.1016/s0272-5231(05)70060-5. PMID 11787659
- [Background] Fiorina C, Vizzardi E, Lorusso R, Maggio M, De Cicco G, Nodari S, Faggiano P, Dei Cas L. The 6-min walking test early after cardiac surgery. Reference values and the effects of rehabilitation programme. Eur J Cardiothorac Surg. 2007 Nov;32(5):724-9. doi: 10.1016/j.ejcts.2007.08.013. Epub 2007 Sep 18. PMID 17881241
- [Background] O'Driscoll BR, Howard LS, Davison AG; British Thoracic Society. BTS guideline for emergency oxygen use in adult patients. Thorax. 2008 Oct;63 Suppl 6:vi1-68. doi: 10.1136/thx.2008.102947. No abstract available. PMID 18838559